CLINICAL TRIAL: NCT01249209
Title: Qualitative Retrospective Study Where the Intervention Consisted of Group Therapy and Individual Interviews Over a Two-year Period
Brief Title: Outpatient Treatment of Patients With Morbid Obesity - a Two-year Follow up
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sykehuset Innlandet HF (Other)
Responsible Party: Sykehuset Innlandet HF, Sykehuset Innlandet HF
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: SI HF Kongsvinger; skyrud,randi (Other: SykehusetInnlandet)
Record Dates: First submitted 2010-11-24; First posted 2010-11-29 (Estimated); Last update posted 2010-11-29 (Estimated); Status verified 2010-06

CONDITIONS: Morbid Obesity
Keywords: obesity; adults; lifestyle intervention; effect after two years treatment for lifestyle change - morbid obesity adults
MeSH Terms: conditions — Obesity, Morbid; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- lifestyle advice (Other)
  Interventions: Device: lifestyle advice

INTERVENTIONS:
Device: lifestyle advice

SUMMARY:
This study is a pilot project to investigate any effect on these markers in conjunction with lifestyle changes / conservative treatment. Useful and significant information in this pilot project is intended to be used as background for further research on this issue in connection with a doctorate.

What is the effect of two years of outpatient treatment for lifestyle change for weight markers, waist, BMI, HbA1c, HDL and LDL cholesterol, triglycerides and uric acid in adults with morbid obesity?

ELIGIBILITY:
Inclusion Criteria:

* Adults from 18 - 60 years, both sex

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2010-05; Primary Completion 2010-09 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Sykehuset Innlandet Kongsvinger, Kongsvinger, Norway